CLINICAL TRIAL: NCT06786156
Title: The Effect of Fetal Movement Counting Given with Pecha Kucha Education on Prenatal Bonding and Pregnancy Distress in Pregnant Women with Placenta Previa
Brief Title: Pregnant Women with Placenta Previa
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, principal investigator midwife, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 08.01.2025/01/26decision no
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Placental Previa
Keywords: Fetal Movement; Pecha Kucha; Pregnancy Distress; Placental Previa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention)
- INTERVENTION 1 (Experimental): Pecha Kucha Education
  Interventions: Behavioral: Pecha Kucha Education

INTERVENTIONS:
Behavioral: Pecha Kucha Education — After the first interviews, the participants will be given face-to-face training to count fetal movements in the first stage. The training will last 30-45 minutes. The training content includes a comfortable environment and a suitable position for pregnant women, how to count and what to look for before counting fetal movements. Then, the training will be sent to the pregnant women via WhatsApp. A form will be given to count the fetal movements, and training will be applied using the Pecha Kucha method using smartphones once a week for 4 weeks. Pecha kucha is a presentation method developed to attract and maintain the attention of the audience throughout a series of different presentations. Pecha kucha (P-K), derived from the word meaning "chat" in Japanese, is to help present creative works with visual images. Pecha kucha training includes position, how to count and what to look for before counting fetal movements. This training will be delivered via WhatsApp with a practical presenta
  Arms: INTERVENTION 1

SUMMARY:
Placenta previa is the extension of placental tissue over the endocervical os or covering the cervical os. Placenta previa is a common complication in the third trimester of pregnancy and is a major cause of postpartum hemorrhage and perinatal death.There are many studies in the literature on attachment. However, no studies have been found on fetal movement in placenta previa pregnant women. Counting fetal movements is an easy and inexpensive assessment that pregnant women can do on their own, without the need for any specialist or equipment, and for which they take responsibility. It is assumed that the effective time spent during fetal movement counting will positively affect the attachment between the pregnant woman and the fetus, and that the stress of the pregnant woman, who is sure that her baby is well, will decrease.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45

  * In the second trimester,
  * Primiparous,
  * With adequate communication skills
  * Literate,
  * Able to read and understand Turkish,

Exclusion Criteria:

Having any mental illness

* Having communication, hearing or vision problems that prevent you from answering the data collection tools

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Prenatal attachment scale | aseline and 3 months.
Tilburg pregnancy distress scale | aseline and 3 months.